CLINICAL TRIAL: NCT01270633
Title: A Multi-Center, Prospective, Randomized Study With Primatrix Dermal Repair Scaffold For The Treatment Of Diabetic Foot Ulcers
Brief Title: A Study With Primatrix Dermal Repair Scaffold For The Treatment Of Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEI-004
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Other): PriMatrix applied to appropriately debrided wound bed and covered with a non-adherent dressing. Dressings applied to maintain moist wound therapy.
  Interventions: Device: PriMatrix
- Standard of Care (Active Comparator): Non adherent dressing applied to appropriately debrided wound bed and moist wound therapy maintained.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: PriMatrix — Following sharp debridement, application of PriMatrix dermal repair scaffold in conjunction with moist wound therapy
  Arms: Treatment
Other: Standard of Care — Following sharp debridement, moist wound therapy
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to compare the clinical and economic effectiveness of PriMatrix and Standard of Care in the treatment of diabetic foot ulcers (DFUs) in subjects with controlled diabetes mellitus and without significantly compromised arterial circulation.

DETAILED DESCRIPTION:
Subjects will be considered for screening upon meeting initial eligibility criteria. After a 2 week screening period, subject will be randomized and enrolled if additional criteria is met. In particular, if wound size has decreased by greater than 40%, subject will be considered a screen fail and randomization will not take place. If all criteria including wound size at Week 3 is met, subject will be randomized and enrolled. Subjects will return weekly for a maximum of 12 weeks, or whenever healing occurs and then once more for a confirmation of healing. Week 24 will consist of a phone call to the subject to complete QOL surveys.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age and able to give their own consent
* Type I or Type II diabetes with investigator-confirmed reasonable metabolic control
* Study ulcer has a Wagner grade of 1 or 2
* Study ulcer size of at least 1 cm2, but not exceeding 20 cm2 in area after debridement
* A full thickness diabetic foot ulcer located on the foot or ankle
* An ulcer which has been in existence for a minimum of 30 days, prior to the day of screening.

Exclusion Criteria:

* Suspected or confirmed signs/symptoms of wound infection
* Wounds with exposed bone or tendon
* Hypersensitivity to bovine collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percent of study ulcers healed | 12 weeks post-randomization
  Percent of study ulcers healed at week 12 post-randomization

SECONDARY OUTCOMES:
Cost of Treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yiannis Monovoukas, PhD, Study Chair — TEI
Locations (8):
- United States (2):
  - HyperbaRXs, Cumming, Georgia
  - Covenant Medical Center, Saginaw, Michigan
- Puerto Rico (6):
  - Caribbean Clinical Trials, San Juan, PR
  - Professional Hospital, Guaynabo
  - Dr. Pila Metropolitan Hospital Wound Healing Center, Ponce
  - Doctors' Center Hospital of San Juan, San Juan
  - Wound and Ulcer Care Clinic of San Juan, San Juan
  - Wilma N. Vazquez Hospital, Vega Baja